CLINICAL TRIAL: NCT04311515
Title: A Phase 2A Study to Evaluate Safety, Tolerability and Pharmacological Effects of PU AD in Subjects With Mild Alzheimer's Disease (AD) Dementia
Brief Title: To Evaluate Safety, Tolerability and Pharmacological Effects of PU AD in Subjects With Mild AD Dementia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Samus Therapeutics company closure
Sponsor: Samus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PU-AD-SD-0201
Record Dates: First submitted 2020-03-12; First posted 2020-03-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy; SyrSpend

STUDY DESIGN:
Intervention Model Description: randomized, double blind, placebo controlled, parallel phase 2a
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All subjects, investigators, and study site personnel will be blinded to dose assignment.
  The Data Safety Monitoring Board (DSMB) will have access to unblinded safety data and will conduct review of these data at regular intervals during the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 30 mg PU AD (Active Comparator): 75 subjects will be treated with active PU-AD on a 1:1 ratio qd
  Interventions: Radiation: Tau Positron emission tomography (PET); Radiation: Fluorodeoxyglucose (FDG) Positron emission tomography (PET); Diagnostic Test: Cerebrospinal fluid (CSF) Biomarkers; Diagnostic Test: Blood Biomarkers; Behavioral: Rating Scales; Drug: PU-AD
- 30 mg Placebo (Placebo Comparator): 75 subjects will be treated with placebo SyrSpend on a 1:1 ratio qd
  Interventions: Radiation: Tau Positron emission tomography (PET); Radiation: Fluorodeoxyglucose (FDG) Positron emission tomography (PET); Diagnostic Test: Cerebrospinal fluid (CSF) Biomarkers; Diagnostic Test: Blood Biomarkers; Behavioral: Rating Scales; Drug: Placebo

INTERVENTIONS:
Radiation: Tau Positron emission tomography (PET) — Tau PET imaging enables the longitudinal assessment of the spatial pattern of tau deposition. Tau accumulates with progression of AD dementia and may be sensitive to disease related changes, particularly those due to intervention with a drug thought to work through a tau related mechanism. Quantitative assessments will be utilized to evaluate the target engagement and pharmacological effects of PU-AD after 6 months of treatment
Radiation: Fluorodeoxyglucose (FDG) Positron emission tomography (PET) — Measurement of neuronal function with FDG PET can help to understand the relationship between target engagement and potential clinical effects. FDG PET will be acquired using stringent quality control. Since glucose metabolism captures all neuronal activity, in order to isolate effects due to treatment, patients will be maintained in a consistent state during the tracer uptake period. Subject motion during image acquisition will be minimized and monitored. Images will be quality controlled, processed, and measured quantitatively using methods that maximize signal to noise associated with technical and physiologic variability
Diagnostic Test: Cerebrospinal fluid (CSF) Biomarkers — A broad set of biomarkers are being assessed in this study to indicate whether this treatment is able to impact multiple pathways associated with AD related to neurodegeneration
Diagnostic Test: Blood Biomarkers — Changes in blood biomarkers may be observable if treatment affects cerebral amyloidosis and loss of nerve cells
Behavioral: Rating Scales — Alzheimer's Disease composite score (ADCOMS+), CDR sb, Alzheimer's Disease Assessment Scale Cognitive (ADAS cog), Alzheimer's Disease Cooperative Study Activities of Daily Living (ADCS ADL), Mini Mental State Examination (MMSE), Alzheimer's Disease Assessment Scale Cognitive (ADAS-COG 12)
Drug: PU-AD — PU-AD 30mg daily for 6mos
  Arms: 30 mg PU AD
Drug: Placebo — Placebo 30mg daily for 6mos
  Other Names: SyrSpend
  Arms: 30 mg Placebo

SUMMARY:
The study is designed as a classic, randomized, double blind, placebo controlled, parallel group study including one active dose of PU AD and matching placebo, designed to assess safety, tolerability and pharmacological effects of oral PU AD (dihydrochloride salt) in subjects with mild AD

DETAILED DESCRIPTION:
This is a multicenter, randomized, double blind, placebo controlled, parallel group Phase 2A study with one active dose of PU AD and matching placebo, once daily (qd), designed to assess safety, tolerability and pharmacological effects of oral PU AD (dihydrochloride salt) in subjects with mild AD. This study will be performed at up to 50 clinical sites in the US and approximately 150 subjects are expected to participate in this study, with 75 subjects in each treatment arm randomized 1:1. Subjects with mild AD meeting all inclusion criteria and none of the exclusion criteria are eligible to participate in this study.

The study consists of a Screening Period (including Pre treatment) (4 weeks), Treatment Period (24 weeks), and a safety Follow up visit (within 30 days [±7 days] after the last dose of IMP). The expected study duration is 24 Months.

The Screening Visit and Pre treatment Visit will take place within 4 weeks of dosing to assess eligibility of subjects. Enrolled subjects will return to the site for randomization and baseline assessments at Week 1. Subjects will be randomized with a 1:1 ratio to one of two treatment arms: 30 mg PU AD or matching 30 mg placebo qd. During the 24 Week Treatment Period, subjects will be administered 30 mg PU AD or matching 30 mg placebo qd, orally. According to investigator's clinical judgement, subjects experiencing intolerable AEs, if medically necessary, may be allowed to adjust the dose regimen from 30 mg qd to 30 mg every other day (qod), with approval by the medical monitor. If patients still cannot tolerate the adjusted dose regimen, the investigator must discuss early termination with the medical monitor.

Subjects will return to the site at Week 2, Week 4, Week 6, Week 12, Week 18, and Week 24 for study assessments as specified PK sampling time points are specified in and will support a population PK model. . Any subject who discontinues prior to completion of the study, and reached 12 weeks of treatment should have all scheduled assessments of the Week 24/Early Termination (ET) Visit completed. All subjects will return to the site for a Follow up Visit, within 30 days (±7 days) after the last dose of study for safety assessments at the Week 28/End of Study (EoS) Visit

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 55 to 80 years old (inclusive)
2. Diagnosis of probable AD dementia based on National Institute on Aging and Alzheimer's Association (NIA/AA) AD Dementia diagnostic criteria
3. Mild AD as assessed by Mini Mental State Examination (MMSE) score between 18 to 26 at Screening Visit (inclusive)
4. Tau positive as evaluated by Tau PET using 18F-PI-2620 and assessment of tracer uptake in the medial temporal lobe and any cortical regions associated with Alzheimer's disease.
5. Geriatric Depression Scale score of ≤ 6 (on the staff administered short form)
6. Magnetic resonance imaging (MRI) or computerized tomography (CT) scan performed within the past 2 years that has confirmed no findings inconsistent with a diagnosis of AD
7. Subjects or his/her caregiver and/or legally authorized representative must have signed and dated an Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written Informed Consent Form (ICF)
8. Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, and other requirements of the study
9. Must have one caregiver who, in the investigator's judgment, has frequent and sufficient contact with the subject (at least 10 hours/week) and is able to provide accurate information about the subject's cognitive and functional abilities; the caregiver must agree to, accompany the subject to clinic visits and/or be available by phone at designated times to provide information to the investigator and study staff about the subject, attend in person clinic visits that require partner input for scale completion, and must agree to monitor the subject's administration of any prescribed medications
10. Female must either be post menopausal (no menstrual period for >1 year), or surgically sterilized (by hysterectomy, bilateral oophorectomy, or bilateral tubal ligation).
11. Males who are sexually active and whose partners are females of childbearing potential must agree to use condoms from screening through 90 days after administration of the last dose of IMP; their partners must be willing to use a medically acceptable method of contraception (a barrier method, intrauterine device, or hormonal contraception) from screening through 90 days after administration of the last dose of IMP
12. Must consent to Apolipoprotein E (ApoE) genotyping; the subject's ApoE status may be disclosed to him/her at the investigator's discretion -

Exclusion Criteria:

1. Meets National Institute of Neurological Disorders and Stroke/Association Internationale pour la Recherche et l'Enseignement en Neurosciences (NINDS/AIREN) criteria for vascular dementia
2. Has current serious or unstable illnesses including cardiovascular, hepatic, renal, gastroenterological, respiratory, endocrinologic, neurologic (other than AD), psychiatric, immunologic, or hematologic disease and other conditions that, in the investigator's opinion, could interfere with the analyses of safety and pharmacologic effect in this study; or has a life expectancy of < 2 years
3. Has had a history within the last 5 years of a serious infectious disease affecting the brain or head trauma resulting in protracted loss of consciousness
4. Has a history within the last 5 years of a primary or recurrent malignant disease with the exception of resected cutaneous squamous cell carcinoma in situ, basal cell carcinoma, cervical carcinoma in situ, or in situ prostate cancer with a normal prostate specific antigen post treatment
5. Has a known history of human immunodeficiency virus (HIV), clinically significant multiple or severe drug allergies, or severe post treatment hypersensitivity reactions
6. Has a "yes" answer to Columbia Suicide Severity Rating Scale (C-SSRS) suicidal ideation item 4 or 5, or any suicidal behavior assessment within 6 months of Screening, or has been hospitalized or treated for suicidal behavior in the past 5 years before Screening
7. Has received acetylcholinesterase inhibitor (AChEIs), memantine, and/or other AD therapy for less than 4 months or has less than 2 months of stable therapy on these treatments
8. Has not been stable on medications that affect the Central nervous system (CNS), for at least 4 weeks (including antidepressants, hypnotics, antipsychotics, etc.) except occasional use of benzodiazepine (definition of occasional use - not more than twice in a week or three times in a month during the past 3 months).
9. Has a history of chronic alcohol or drug abuse/dependence within the past 5 years
10. Any medical or neurological/neurodegenerative condition (other than AD) that, in the opinion of the investigator, might be a contributing cause to the subject's cognitive impairment (e.g., current history of substance abuse, uncontrolled vitamin B12 deficiency or abnormal thyroid function, stroke or other cerebrovascular condition, Parkinson's disease, Lewy body dementia, or frontotemporal dementia)
11. Transient ischemic attack or stroke or any unexplained loss of consciousness within 1 year prior to Screening Visit
12. History of bleeding disorder or predisposing conditions, blood clotting, or clinically significant abnormal results on coagulation profile at Screening, as determined by the investigator
13. History of unstable angina, myocardial infarction, chronic heart failure (New York Heart Association Class III or IV), or clinically significant conduction abnormalities (e.g., unstable atrial fibrillation) within 1 year prior to Screening Visit
14. Clinically significant 12 lead Electrocardiogram (ECG) abnormalities, as determined by the investigator
15. Indication of impaired liver function as shown by an abnormal liver function profile at Screening (e.g., repeated values of Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≥ 2 × the upper limit of normal [ULN]) and/or indication of impaired renal function at Screening (e.g., repeated values of creatinine and blood urea nitrogen [BUN] ≥ 1.5 × Upper limit of normal (ULN) or estimated glomerular filtration rate < 45 mL/minute/1.73 m2 and corroborating medical history and physical examination)
16. Contraindications to having a brain Magnetic resonance imaging (MRI) (e.g., MRI incompatible pacemaker; MRI incompatible aneurysm clips, artificial heart valves, or other metal foreign body; claustrophobia that cannot be medically managed); if the MRI compatibility of implanted devices is unknown, the subject must be excluded from the study
17. Contraindication to having a PET brain scan (e.g., inability to lie flat or still for the duration of the scan) or intolerance to previous PET scans (i.e., previous hypersensitivity reactions to any PET ligand or imaging agent, failure to participate in and comply with previous PET scans)
18. Contraindication to having an FDG PET scan, including uncontrollable glucose levels, inability to fast for the prescribed number of hours prior to the FDG PET scan, inability to withhold all insulin and oral diabetic medication after midnight prior to the PET scan
19. Inability to refrain from using sleep medication for the 24 hours prior to each FDG PET scan or to refrain from use of antipsychotics, sedatives, or other strong acting neuropsychiatric medication on the day of each PET scan prior to the scan
20. Current or recent participation (within 12 months before screening) in any procedures involving radioactive agents such that radiation exposure of the, in the judgement of the investigator (upon review of medical history), subject in any given year would exceed the whole-body limits of annual and total dose commitment of 5 rems set forth in the US Code of Federal Regulations (CFR) Title 21 section 361.1.
21. Any contraindications to lumbar puncture (LP), e.g., increased bleeding risk (platelet count <100,000/μL, coagulopathies, anticoagulant drugs), lumbar spine deformity that might interfere with the procedure evidence on MRI contraindicating LP, risk for cerebral herniation, space occupying lesion with mass effect, abnormal intracranial pressure due to increased CSF pressure, Arnold Chiari malformation, local infections at the puncture site and patient fear of LP; abnormalities in the screening CSF profile that are considered by the Investigator to be clinically significant are exclusionary
22. Any major surgery within 12 weeks of Screening Visit or during the Screening Period
23. Has active ocular condition that in the opinion of the investigator may alter visual acuity during the course of the study.
24. Use of any drugs that are strong inhibitors of Cytochrome (CYP)450 (2D6 or 2C19) within 7 days or 5 half lives of the inhibitor (whichever is longer), prior to administration of the first dose of Investigational medicinal product (IMP) and/or plan to use throughout the study
25. Participation within the 12 months prior to Screening Visit in a study of any agent(s) with a purported disease modifying effect in AD (e.g., anti beta amyloid, β secretase inhibitors, γ secretase inhibitors), unless documentation of receipt of placebo is available
26. Has taken other investigational drugs or participated in any clinical study within 30 days or 5 half lives (if known) of the investigational drug, whichever is longer, prior to first dose of IMP in this study or is currently participating in another clinical study
27. Other unspecified reasons that, in the opinion of the investigator or Samus, and/or its delegated medical monitor, make the subject unsuitable for the study

    -

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Fluorodeoxyglucose Positron emission tomography (FDG-PET) | 6 months
  Change from baseline in pharmacologic parameters over 6 months for FDG-PET measurements
incidence and severity of Adverse Events (AEs), serious adverse events (SAEs) | 6 months
  safety and tolerability, assessed by incidence and severity of AEs, SAEs, and AE's leading to withdrawal of treatment during the course of the study

SECONDARY OUTCOMES:
Tau Positron emission tomography (Tau PET )standardized uptake value ratio (SUVR) | 6 months
  Change from baseline in pharmacologic parameters over 6 months measurements
Ratio of p-Tau to t-tau in Cerebrospinal fluid (CSF) | 6 months
  Change from baseline in pharmacologic parameters over 6 months using Ratio of p-Tau to t-tau in Cerebrospinal fluid (CSF)
Alzheimer's Disease composite score (ADCOMS) | 6 months
  Change from baseline in pharmacologic parameters over 6 months using ADCOMS scales
Global Statistical Test (GST) combining Alzheimer's Disease Assessment Scale Cognitive (ADAS-Cog), Alzheimer's Disease Cooperative Study Activities of Daily Living (ADCS-ADL), and Clinical Dementia Rating Sum of Boxes (CDR-sb) | 6 months
  Change from baseline in pharmacologic parameters over 6 months using Global Statistical Test (GST) combining Alzheimer's Disease Assessment Scale Cognitive (ADAS-Cog), Alzheimer's Disease Cooperative Study Activities of Daily Living (ADCS-ADL), and Clinical Dementia Rating Sum of Boxes (CDR-sb)
Pharmacokinetic (PK) | 6 months
  PK of PU-AD in this population

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Silverman, MD, Study Director — Samus Therapeutics Consultant
Locations (10):
- United States (10):
  - SFM Clinical Research, LLC, Boca Raton, Florida
  - Brain Matters Research, Delray Beach, Florida
  - JEM Research, Lake Worth, Florida
  - Med-Care Research, Miami, Florida
  - Miami Dade Medical Research Institute, LLC, Miami, Florida
  - Neurostudies, Inc, Port Charlotte, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Conquest Research LLC, Winter Park, Florida
  - Advanced Clinical Institute, Inc., Neptune City, New Jersey
  - Princeton Medical Institute, Princeton, New Jersey

IPD SHARING:
Plan to Share IPD: No